

## Statistical Analysis Plan

## **Study Title:**

To investigate the potential effectiveness of mirror-aided cross-education using the innovative 'Mirror Strengthening Device' compared to mirror therapy alone in post-stroke upper limb recovery: A pilot randomised feasibility study.

**Document creation date:** February 4<sup>th</sup> 2022

NCT number [not yet assigned].

Identifiers: [NCT ID not yet assigned]



## **Statistical Analysis**

We will analyse the data using Excel and SPSS for Windows. Paired T tests will be used to compare before and after data in both groups.